CLINICAL TRIAL: NCT03843840
Title: Combined Coaxial Optical Coherence Tomography System to Image the Retina and Choroidal Structures and Estimate Tissue Reflectivity in Healthy and Diseased Retinas
Brief Title: Dual Wavelength OCT
Status: Completed | Type: Observational
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: TUFA1040
Record Dates: First submitted 2018-05-31; First posted 2019-02-18 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: AMD; Diabetic Retinopathy; Retinal Degeneration; Retinal Dystrophies
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Degeneration; Retinal Dystrophies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diseased Retina
  Interventions: Device: Combined Coaxial Optical Coherence Tomography

INTERVENTIONS:
Device: Combined Coaxial Optical Coherence Tomography — Taking images of the retina with two wavelengths

SUMMARY:
The purpose of this research is the evaluation of a combined coaxial optical coherence tomography (OCT) system to image retina/choroid and to evaluate if post processing of the data can give us insights into property of the tissue imaged.

DETAILED DESCRIPTION:
Histology studies have shown that many disorders of the retina and choroid such as age-related macular degeneration is associated with a build up abnormal deposits, in the retina or subretinal space. Being able to detect subtle changes in retina and choroidal structure is crucial for better understanding and monitoring of this potentially blinding condition. This study aims to commercially available Spectralis® OCT-system with a central wavelength of 880nm explore the ability of a confocal scanning laser ophthalmoscope (cSLO) for OCT imaging utilising a modified by the addition of a longer wavelength OCT (1075nm , a wavelength deployed on other commercially available OCT scanners). Other commercially available OCT scanners used longer wavelengths to allow deeper penetration and enhanced visualisation of subretinal tissue but less inner retinal detail. Combing both wavelengths could have the advantage of allowing optimum viualisation of inner and subretinal structures. The ability of the systems to acquire repeatable and good quality images of retinal and choroidal structural detail at matching location and compare the results from the two instruments will be evaluated. In addition processing of the images reflectivity with two different wavelength should give us insight into the nature of any abnormal material.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* Ability to consent
* Abnormal reflectivity detected in at least one eye in the retina or choroid on OCT testing undertaken as part of routine
* clinical care

Exclusion Criteria:

* Media opacities on conventional OCT testing taken on the day of the study visit, that prevents adequate visualisation of
* the retina and/or choroidal substructures in the opinion of the investigator
* Inability to undertake to undertake two additional OCT scans on each eye in addition to their conventional OCT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with diseased retina
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Test retest reliability | 14 months
  Comparison of device test retest variability with those of standard OCT for measurement of tissue reflectivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, 162 City Road, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No